CLINICAL TRIAL: NCT01764360
Title: Strategies to Improve Kaposi Sarcoma (KS) Outcomes in Zimbabwe (SIKO)
Brief Title: Strategies to Improve Kaposi Sarcoma (KS) Outcomes in Zimbabwe
Acronym: SIKO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-0816
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Kaposi Sarcoma (KS); HIV
MeSH Terms: conditions — Sarcoma, Kaposi

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- KS structured clinical care training (Other): Eight primary care sites in Zimbabwe will be randomized at different timepoints to receive structured training for diagnosis and treatment of Kaposi sarcoma (KS)
  Interventions: Other: KS structured clinical care training

INTERVENTIONS:
Other: KS structured clinical care training — Eight primary care sites in Zimbabwe will receive structured training for diagnosis and treatment of Kaposi sarcoma (KS)

SUMMARY:
Kaposi sarcoma (KS) is an AIDS-related cancer and is the most commonly reported cancer in Zimbabwe. If it is found early on, it may be treatable with antiretroviral therapy (ARVs) alone and this will improve general well-being and ease of care. It may also be possible to avoid use of expensive chemotherapy if the KS is picked up early on in the course of the disease. Early KS is often overlooked or not recognized by health professionals. The purpose of the study is to learn more about if the level of medical care and treatment provided at primary care clinics in Zimbabwe will help people with AIDS-KS do better and maintain their health longer. This will be done by monitoring how KS is diagnosed and treated at the primary care clinics. Clinics will then have training in how to recognize and treat KS so that they can better identify and care for patients with the disease.

DETAILED DESCRIPTION:
The "Strategies to Improve Kaposi Sarcoma (KS) Outcomes in Zimbabwe" (SIKO Study) will consist of both an interventional and an observational component. Eight (8) primary care sites in Zimbabwe will be randomized to receive structured training on Kaposi sarcoma (KS) diagnosis and treatment. This intervention will be evaluated through the utilization of three components; the KS Standardized Evaluation (KS-SE), integration of palliative care and an algorithm-based KS management strategy at the sites. The impact of the overall intervention will be evaluated using a step-wedge randomized cluster trial design in which the 8 primary care sites will be randomized to receive the intervention at different time points such that the intervention will be eventually be implemented at all sites during the 2 year (102 weeks) course of the study. The 2 year evaluation period will consist of a monitoring period, followed by an intervention period.

The observational component of the SIKO study will be the enrollment of all patients who are found to have Kaposi sarcoma (KS) during either the monitoring or intervention periods at any of eight study sites. After informed consent is obtained, information of HIV status, KS diagnosis and staging, demographic data and a quality of life questionnaire will be collected, along with A glycoprotein predominantly found on the surface of helper T cells. (CD4+) counts (if available), antiretroviral (ARV) medication and tuberculosis and KS treatment history. Patients will continue to be followed over the course of the study.

For power estimations we assumed each site would enroll between 0·5 to 0·7 subjects per week, resulting in final sample sizes of 158 to 221 in the Pre-Intervention Period and 318 to 445 in the Intervention Period. To evaluate the effect of the Intervention Package on T0 (T0/(T0 + T1)) we assumed T0 proportions of 0·12 to 0·15 during the Pre-Intervention Period, within site correlations of 0·10, 0·15 and 0·20, and a maximum enrollment of 100 per site. We estimated 80% power to detect a minimum increase of the T0 proportion from 0·12 to 0·37 or from 0·15 to 0·40. Power estimation for evaluation of time to loss-to-care assumed a Kaplan-Meier approach and provided 80% power to detect a hazard ratio (HR) ≥ 1·89 with a total sample of up to 512 KS cases. Sample sizes were calculated using PASS, (NCSS software, Kayesville UT), assuming a 0·05 two-sided significance level.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 1 and 80,
* Recruited from the eight (8) participating primary care sites,
* Subjects newly identified with Kaposi sarcoma (KS) and HIV-1 infection.

Exclusion Criteria:

* None Noted

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1024 (Actual)
Dates: Start 2013-02; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in identification of early stage diagnosis of Kaposi Sarcoma (KS) | 2 years
  Compare the proportions of new KS diagnoses identified as Stage T0 (early stage) during the standard-of-care and the SIKO intervention periods.
Change in access to palliative care | 2 years
  Compare the Functional Living Index-Cancer (FLI-C) quality-of-life score in evaluating physical and emotional symptom distress during the standard-of-care and the SIKO intervention periods.
Change in survival and retention in care | 2 years
  Evaluate the events (failure to attend clinic, refill prescriptions; to include both death and non-death causes of loss of care) leading to non-retention in care. Compare time to loss of care for all new AIDS-KS patients diagnosed during the standard-of-care and the SIKO intervention periods.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B. Campbell, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Zimbabwe College of Health Sciences, Harare, Zimbabwe

REFERENCES:
- [Derived] Sabourin KR, Borok M, Mawhinney S, Matimba M, Jaji F, Fiorillo S, Chifamba DD, Muserere C, Mashiri B, Bhodheni C, Gambiza P, Mandidewa R, Mutimuri M, Gudza I, Mulvahill M, Moore CM, Kutner JS, Simoes EAF, Campbell TB. Evaluation of a training intervention to improve cancer care in Zimbabwe: Strategies to Improve Kaposi Sarcoma Outcomes (SIKO), a prospective community-based stepped-wedge cluster randomized trial. J Int AIDS Soc. 2022 Aug;25(8):e25998. doi: 10.1002/jia2.25998. PMID 36028920